CLINICAL TRIAL: NCT00996333
Title: Phase II Study of a Biochemically Synergistic Regimen for Metastatic Pancreatic Cancer (Stage IVB) With Gemzar, Taxotere and Xeloda (GTX)
Brief Title: Study of Gemzar®, Taxotere®, and Xeloda® (GTX) in Patients With Metastatic Pancreatic Cancer (Stage IVB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB8628
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Stage IVB
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemzar, Taxotere, Xeloda (Experimental): Gemcitabine, Docetaxel, Capecitabine:
  Gemzar intravenously on Day 4 and 11 Taxotere intravenously on Day 4 and 11 Xeloda tablet taken orally every day for 14 days
  Interventions: Drug: Gemcitabine, Docetaxel, Capecitabine

INTERVENTIONS:
Drug: Gemcitabine, Docetaxel, Capecitabine — 1500mg/m2/day of Capecitabine for 14 days 750mg/m2 of Gemcitabine on Day 4 and 11 30mg/m2 of Docetaxel on Day 4 and 11
  This 2-week regimen is followed by 1 week off for a total of a 21-day cycle. This is repeated for a total of 3 cycles.
  Other Names: Gemzar; Xeloda; Taxotere

SUMMARY:
This study is designed to determine whether an investigational drug combination consisting of Gemzar®, Taxotere®, and Xeloda®, (called GTX) is safe and effective in treating advanced pancreatic cancer and to study and enhance the utility of PET scans in the evaluation of patients with pancreatic cancer.

DETAILED DESCRIPTION:
This Phase II multicenter study is designed to determine the response rate to a biochemically synergistic regimen with Gemzar, Taxotere, and Xeloda in patients with Stage IVB metastatic pancreatic cancer. It will further determine the overall and one year survival rates, the diseasefree interval, and the toxicities for this regimen in patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of pancreas metastatic to liver and/or lungs or peritoneal surface. (a.k.a. Stage IV B).
* No prior chemotherapy with Gemzar, Xeloda and Taxotere.
* Measurable disease: Any mass reproducibly measurable in two perpendicular diameters by x-ray, physical examination, CT or MRI scans.
* The following lesions conventionally are not considered measurable:

  * CNS lesions
  * Blastic or lytic bone lesions (which should be documented and followed)
  * Radiated lesions unless progression after RT is documented
* Ineligible for other high priority national or institutional studies
* Prior radiation and surgery allowed:

  * > 3 weeks since surgery
  * > 4 weeks since RT
* Non pregnant females who are not breast feeding with a negative serum or urine β-HCG test within 1 week of starting the study. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter.
* Clinical Parameters:

  * Life expectancy > 2 months
  * Age 18 - 70 years old
  * Performance status 0-2 (ECOG)
  * Peripheral Neuropathy must be < grade 1
  * Able to tolerate oral medications
* Required initial laboratory data:

  * Absolute Neutrophil Count > 1,500 μl
  * White Blood Count > 3,000/μl
  * Platelet count > 100,000/μl
  * BUN < 1.5 x normal
  * Creatinine < 1.5 normal
  * Hemoglobin > 8.0 g/dl
  * Serum Albumin > 3 mg/dl
  * Total Bilirubin < 2.0 mg/dl
  * SGOT, SGPT, Alkaline Phosphatase SGOT and SGPT may be up to 3.0 x ULN if Alk Phos < 2.0 x ULN; or Alk Phos may be up to 3.0 x ULN if SGOT and SGPT are < 2.0 x ULN

Exclusion Criteria:

* Hypersensitivity: Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80 must be excluded.
* Informed Consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.
* The patient has not had a prior malignancy in last 5 years other than curatively treated carcinoma in-situ of the cervix or non-melanoma skin cancer
* No serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g., serious infection).
* Patients with brain metastases are excluded.
* Patients known to have HIV will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Fine, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemzar, Taxotere, Xeloda: Gemzar intravenously on Day 4 and 11 Taxotere intravenously on Day 4 and 11 Xeloda tablet taken orally every day for 14 days
  Gemcitabine, Docetaxel, Capecitabine: 1500mg/m2/day of Capecitabine for 14 days 750mg/m2 of Gemcitabine on Day 4 and 11 30mg/m2 of Docetaxel on Day 4 and 11
  This 2-week regimen is followed by 1 week off for a total of a 21-day cycle. This is repeated for a total of 3 cycles.
Period: Overall Study
Arm/Group | Gemzar, Taxotere, Xeloda
Started | 46
Completed | 33
Not Completed | 13
Not completed — Screen failure | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 4
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Gemzar, Taxotere, Xeloda
Number analyzed (Participants) | 46
Age, Customized [Number; unit: participants]
  Between 30 and 39 years | 2
  Between 40 and 49 years | 4
  Between 50 and 59 years | 16
  Between 60 and 69 years | 20
  Between 70 and 79 years | 3
  Unknown | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: To Determine Response Rate to the GTX Regimen in Patients With Pancreatic Cancer
Description: Data was not analyzed because original PI left institution before data analysis was completed.
Time Frame: 10 weeks
Arm/Group | Gemzar, Taxotere, Xeloda
Number analyzed (Participants) | 0

2. Secondary Outcome: Determine Overall and One Year Survival Rates
Description: Data was not analyzed because original PI left institution before data analysis was completed.
Time Frame: One year
Arm/Group | Gemzar, Taxotere, Xeloda
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity Assessment
Description: Data was not analyzed because original PI left institution before data analysis was completed.
Time Frame: Every month
Arm/Group | Gemzar, Taxotere, Xeloda
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: AE data was only collected on 45 subjects (out of 46 subjects, 1 was a screen failure).
Groups:
- Gemzar, Taxotere, Xeloda: Gemcitabine, Docetaxel, Capecitabine:
  Gemzar intravenously on Day 4 and 11 Taxotere intravenously on Day 4 and 11 Xeloda tablet taken orally every day for 14 days
  Gemcitabine, Docetaxel, Capecitabine: 1500mg/m2/day of Capecitabine for 14 days 750mg/m2 of Gemcitabine on Day 4 and 11 30mg/m2 of Docetaxel on Day 4 and 11
  This 2-week regimen is followed by 1 week off for a total of a 21-day cycle. This is repeated for a total of 3 cycles.
Arm/Group | Gemzar, Taxotere, Xeloda
Serious Adverse Events (participants affected / at risk) | 16/45
Other Adverse Events (participants affected / at risk) | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemzar, Taxotere, Xeloda (N=45)
Surgery (Surgical and medical procedures) | 1 (1)
Alveolitis leading to death (General disorders) | 1 (1)
Leg edema (General disorders) | 1 (1) — Hospitalized
Fever and chills (General disorders) | 2 (2) — Hospitalized
Fever and infection (Infections and infestations) | 1 (1) — Hospitalized
Headache (General disorders) | 1 (1) — Hospitalized
Temporary loss of vision in the right eye (Eye disorders) | 1 (1) — Hospitalized
Small bowel (Gastrointestinal disorders) | 1 (1) — Hospitalized
Pancytopenia and diarrhea (Blood and lymphatic system disorders) | 1 (1) — Hospitalized
Lower abdominal and back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Hospitalized
Leukopenia and hypotension (Blood and lymphatic system disorders) | 1 (1) — Hospitalized
Sepsis and neutropenia (Infections and infestations) | 1 (1) — Hospitalized
Mucositis (Gastrointestinal disorders) | 1 (1) — Hospitalized
Port-a-cath (Surgical and medical procedures) | 1 (1)
Shortness of breath (General disorders) | 1 (1) — Hospitalized
Blood clot (Vascular disorders) | 1 (1) — Hospitalized
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Hospitalized
Constipation, nausea and vomiting (General disorders) | 1 (1) — Hospitalized
Hyponatremia and elevated liver enzymes (Hepatobiliary disorders) | 1 (1) — Hospitalized for this event. Also suffered from dilation of small bowel with pneumatosis.
Death due to unknown reason (General disorders) | 2 (2)
Heart attack leading to death (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemzar, Taxotere, Xeloda (N=45)
Vomiting (General disorders) | 1 (1)
Syncope (Vascular disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes